CLINICAL TRIAL: NCT03489330
Title: A Retrospective Study to Understand the Risk Factors/Drivers of "Inappropriate" Antimicrobial Use and the Performance Evaluation of a Clinical Decision Support Tool That Facilitates Prediction of Outbreaks of Inappropriate Antibiotic Use
Brief Title: Antibiotic Outbreak, Risk Factors for Never Event, Prediction of Inappropriate Use
Status: Completed | Type: Observational
Sponsor: Midwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other); University of Michigan (Other); Henry Ford Hospital (Other); Wayne State University (Other)
Responsible Party: Sponsor
Other Study IDs: MWU3004_STU00205629
Record Dates: First submitted 2018-03-18; First posted 2018-04-05 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Infectious Disease
Keywords: Anti-Bacterial Agents/therapeutic use; Drug Utilization/statistics & numerical data; Hospitals/statistics & numerical data; Data Analysis, Statistical; Interpretation, Statistical Data; Antibiotic Stewardship; Electronic Medical Record
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Northwestern Memorial Hospital data: Inpatient intravenous vancomycin use
- Henry Ford Hospital data: Inpatient intravenous vancomycin use
- University of Michigan Hospital data: Inpatient intravenous vancomycin use

SUMMARY:
In order to decrease inappropriate antibiotic use, drivers of inappropriate use must be identified locally. This study will focus on the MOST inappropriate use, which are defined as 'never events'. Previous work has shown that antibiotic use clusters over time. It is hypothesized that never events also cluster over time. Using electronic data capture strategies, an algorithm will be developed to quickly and accurately identify areas of antibiotic use concern. Secondly, a framework will be developed, utilizing antimicrobial consumption data and captured signals of inappropriate antimicrobial use to provide targets for antimicrobial stewardship efforts.

DETAILED DESCRIPTION:
Appropriateness in antimicrobial prescribing has become a focal national and international issue. It has been estimated that upwards of 50% of antibiotic use is inappropriate. With this backdrop, a national strategic goal has been set by the United States White House to decrease inappropriate antibiotic use by 20% and 50%, respectively for inpatient and outpatient settings. In order to decrease inappropriate use, drivers of incorrect use must be identified at each local setting. The actual drivers of confirmed inappropriate use have been difficult to identify except when using time and resource intense chart reviews. Even the largest contemporary antibiotic consumption studies have not assessed appropriateness as it was 'outside of study scope'. Further, there is no consensus or agreement on what constitutes inappropriate use. These apparent omissions underscore the difficulty and complexity in attributing appropriateness of use for antimicrobials. Importantly, this study will focus on the MOST inappropriate use, which are defined as 'never events'. Previous work has shown that antibiotic use clusters over time. It is hypothesized that never events also cluster over time. Using electronic data capture strategies, an algorithm will be developed to quickly and accurately identify areas of antibiotic use concern. Secondly, a framework will be developed, utilizing antimicrobial consumption data and captured signals of inappropriate antimicrobial use to provide targets for antimicrobial stewardship efforts.

ELIGIBILITY:
Inclusion Criteria:

* receipt of inpatient intravenous vancomycin during proposed study period
* adults 18 years of age or older and less than 90 years of age

Exclusion Criteria:

* individuals who are not yet adults (infants, children, teenagers)
* pregnant women
* prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The retrospective study population will be based on all inpatient intravenous vancomycin used during the proposed 36-month study period. Patient level data that identifies adults unable to consent, individuals who are not yet adults, pregnant women, or prisoners will not be collected.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
appropriateness of vancomycin use | Proposed 36 month study period
  classified as 1) never event, 2) potentially inappropriate, 3) not inappropriate

SECONDARY OUTCOMES:
outbreaks of never events | Proposed 36 month study period
  predictive interval thresholds that identify high proportion of never events

CONTACTS AND LOCATIONS:
Overall Officials: Marc H Scheetz, PharmD, MSc, Principal Investigator — Midwestern University
Locations (1):
- Midwestern University, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All files containing patient identifiers will be de-identified before sharing across study sites.

REFERENCES:
- [Background] Scheetz MH, Crew PE, Miglis C, Gilbert EM, Sutton SH, O'Donnell JN, Postelnick M, Zembower T, Rhodes NJ. Investigating the Extremes of Antibiotic Use with an Epidemiologic Framework. Antimicrob Agents Chemother. 2016 May 23;60(6):3265-9. doi: 10.1128/AAC.00572-16. Print 2016 Jun. PMID 27001807
- [Background] P.R. Yarnold, R.C. Soltysik, Refining two-group multivariable classification models using univariate optimal discriminant analysis., Decision Sciences, 22 (1991) 1158-1164.
- [Background] P.R. Yarnold, R.C. Soltysik, Maximizing Predictive Accuracy, ODA Books2016.
- [Background] Rhodes NJ, O'Donnell JN, Lizza BD, McLaughlin MM, Esterly JS, Scheetz MH. Tree-Based Models for Predicting Mortality in Gram-Negative Bacteremia: Avoid Putting the CART before the Horse. Antimicrob Agents Chemother. 2015 Nov 23;60(2):838-44. doi: 10.1128/AAC.01564-15. Print 2016 Feb. PMID 26596934
- [Background] Cusini A, Rampini SK, Bansal V, Ledergerber B, Kuster SP, Ruef C, Weber R. Different patterns of inappropriate antimicrobial use in surgical and medical units at a tertiary care hospital in Switzerland: a prevalence survey. PLoS One. 2010 Nov 16;5(11):e14011. doi: 10.1371/journal.pone.0014011. PMID 21103362
- [Background] Glowacki RC, Schwartz DN, Itokazu GS, Wisniewski MF, Kieszkowski P, Weinstein RA. Antibiotic combinations with redundant antimicrobial spectra: clinical epidemiology and pilot intervention of computer-assisted surveillance. Clin Infect Dis. 2003 Jul 1;37(1):59-64. doi: 10.1086/376623. Epub 2003 Jun 23. PMID 12830409
- [Background] Hecker MT, Aron DC, Patel NP, Lehmann MK, Donskey CJ. Unnecessary use of antimicrobials in hospitalized patients: current patterns of misuse with an emphasis on the antianaerobic spectrum of activity. Arch Intern Med. 2003 Apr 28;163(8):972-8. doi: 10.1001/archinte.163.8.972. PMID 12719208
- [Background] Fleming-Dutra KE, Hersh AL, Shapiro DJ, Bartoces M, Enns EA, File TM Jr, Finkelstein JA, Gerber JS, Hyun DY, Linder JA, Lynfield R, Margolis DJ, May LS, Merenstein D, Metlay JP, Newland JG, Piccirillo JF, Roberts RM, Sanchez GV, Suda KJ, Thomas A, Woo TM, Zetts RM, Hicks LA. Prevalence of Inappropriate Antibiotic Prescriptions Among US Ambulatory Care Visits, 2010-2011. JAMA. 2016 May 3;315(17):1864-73. doi: 10.1001/jama.2016.4151. PMID 27139059
- [Background] Kelesidis T, Braykov N, Uslan DZ, Morgan DJ, Gandra S, Johannsson B, Schweizer ML, Weisenberg SA, Young H, Cantey J, Perencevich E, Septimus E, Srinivasan A, Laxminarayan R. Indications and Types of Antibiotic Agents Used in 6 Acute Care Hospitals, 2009-2010: A Pragmatic Retrospective Observational Study. Infect Control Hosp Epidemiol. 2016 Jan;37(1):70-9. doi: 10.1017/ice.2015.226. Epub 2015 Oct 12. PMID 26456803
- [Background] Magill SS, Edwards JR, Beldavs ZG, Dumyati G, Janelle SJ, Kainer MA, Lynfield R, Nadle J, Neuhauser MM, Ray SM, Richards K, Rodriguez R, Thompson DL, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Prevalence of antimicrobial use in US acute care hospitals, May-September 2011. JAMA. 2014 Oct 8;312(14):1438-46. doi: 10.1001/jama.2014.12923. PMID 25291579
- [Background] Baggs J, Fridkin SK, Pollack LA, Srinivasan A, Jernigan JA. Estimating National Trends in Inpatient Antibiotic Use Among US Hospitals From 2006 to 2012. JAMA Intern Med. 2016 Nov 1;176(11):1639-1648. doi: 10.1001/jamainternmed.2016.5651. PMID 27653796
- [Background] Rhodes NJ, Wagner JL, Gilbert EM, Crew PE, Davis SL, Scheetz MH. Days of Therapy and Antimicrobial Days: Similarities and Differences Between Consumption Metrics. Infect Control Hosp Epidemiol. 2016 Aug;37(8):971-973. doi: 10.1017/ice.2016.109. Epub 2016 May 13. PMID 27174570
- [Background] The World Health Organization. Health Topics: Disease Outbreaks, 2015.
- See also: Related Info — https://psnet.ahrq.gov/primers/primer/3/never-events

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03489330/SAP_000.pdf
  • Study Protocol (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03489330/Prot_001.pdf